CLINICAL TRIAL: NCT05441241
Title: Reduction of Pain and Distress in Pediatric Population Undergoing a Venipuncture With Active Production of Music With the Leap Motion Controller - a Randomized Controlled Trial
Brief Title: Leap Motion Controller for Pain During Venipuncture in Pediatrics
Acronym: LeapRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 51/2022
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Procedural Pain; Venipuncture
Keywords: Procedural Pain; Venipuncture; Children, Distraction
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leap Motion Controller (Experimental)
  Interventions: Device: Leap Motion Controller
- Standard care (Active Comparator)
  Interventions: Other: Traditional distraction techniques

INTERVENTIONS:
Device: Leap Motion Controller — The Leap Motion Controller is an infrared device that digitalizes in real-time the movements of the hand above it. This signal will be converted into Musical Instrument Digital Interface (MIDI) and then translated into a sound of a pitch that depends on the distance between the hand and the device. The software is set to produce a pentatonic scale, so every melody created by the patient will sound consonant, and the timbre will be warm, calm and in human vocal range (similar to a cello). The operator will do an example, playing a melody, and will invite the patient to imitate him. When the patient gains confidence with the device, after a limited time lapse (from 30 seconds to 3 minutes), while they are playing it with one hand, the venipuncture is done on the other arm
  Arms: Leap Motion Controller
Other: Traditional distraction techniques — Common distraction techniques will be used (i.e., visual stimulation, lecture)
  Arms: Standard care

SUMMARY:
Venipuncture is the most frequent invasive procedure in hospitals and clinics. In the pediatric population this is very often associated with fear, anxiety, distress and enhanced perception of pain. Local anesthetic creams (like EMLA) are used to reduce pain and distress but they need 30-60 minutes of waiting between the application and the puncture, which is too much time for most of everyday life clinical contests. Many distraction techniques have been studied, both active (ie video games, virtual reality) and passive (ie listening to music, visual stimulation).

Active production of music is one of the most complex activities for our central nervous system. It requires a precise timing of a lot of well-coordinated actions, like recognition and conservation of a rhythmic structure, precise execution of quick and complex fine movements, and with an important involvement of intense emotional experience. It stimulates bilaterally primary and secondary auditory cerebral areas, but also motor and premotor areas, language areas and their contralateral, cognitive areas. At the same time, it activates reward and gratification circuits with stimulation of the limbic system and endorphin release and also neurovegetative system. Music is probably the most immediate and spontaneous communication tool that can also act at subcortical level without the person being aware of what they are receiving and transmitting. Music activates the dopaminergic mesolimbic system, which regulates memory, attention, executive functions, motivation and also mood and pleasure through the nucleus accumbens. It also produces measurable cardiovascular and endocrine responses indicated by reduced serum cortisol levels and inhibition of cardiovascular stress reactions.

The Leap Motion Controller is an infrared device that digitalizes the movements of the hand above it in real-time: this is connected with a software that converts this signal into a musical tone specifically set. The melody is created very easily just by moving the hand above it. With this device, children will be able to produce music without anything interposing between them and the sound production. This will allow the patient to focus only on the melodies, without technical difficulties that could derive for instance from a visual interface or an instrument you have to hold.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8-17 years undergoing venipuncture

Exclusion Criteria:

* Patients with cognitive impairment
* Patients who do not understand the Italian language or with parents who are unable to provide a written informed consent in Italian language
* Patients medicated with local anaesthetic cream

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Difference in procedural pain score between experimental and control group | 1 minutes after the procedure
  Procedural pain self-reported by children using the Faces Pain Scale Revised (FPS-R scale). The FPS-R algometric scale includes both a series of smiley faces with an expression that changes according to increasing pain, and a numerical scale, for a pain scale ranging from zero (no pain) to 10 (severe pain).

SECONDARY OUTCOMES:
Difference in child distress between experimental and control group evaluated by parents | 1 minutes before the procedure
  The distress score will be evaluated by parents through the Distress thermometer, a single-item tool using a 0 (no distress) to 10 (extreme distress)-point Likert scale resembling a thermometer.
Difference in child distress between experimental and control group evaluated by health operators | 1 minutes before the procedure
  The distress score will be evaluated by health operators through the Distress thermometer, a single-item tool using a 0 (no distress) to 10 (extreme distress)-point Likert scale resembling a thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: Egidio Barbi, MD, Principal Investigator — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Obersnel M, Nardin B, Canepari E, Torelli L, Rizzitelli P, Buchini S, Schreiber S, Barbi E, Cozzi G. Active production of music as distraction for venipuncture in children and adolescents: a randomized clinical trial. Eur J Pediatr. 2023 Dec;182(12):5455-5463. doi: 10.1007/s00431-023-05227-2. Epub 2023 Sep 29. PMID 37773297